CLINICAL TRIAL: NCT04550104
Title: A Platform Study of DNA Damage Response Inhibitors in Combination With Conventional Radiotherapy in Non Small Cell Lung Cancer
Brief Title: A Platform Study of Novel Agents in Combination With Radiotherapy in NSCLC
Acronym: CONCORDE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: University of Manchester (Other); Newcastle University (Other); University of Oxford (Other); The Leeds Teaching Hospitals NHS Trust (Other); Beatson West of Scotland Cancer Centre (Unknown); University of Glasgow (Other); Velindre NHS Trust (Other Government); University College London Hospitals (Other); Queen's University, Belfast (Other); University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO20/118073; 2020-000206-28 (EudraCT Number); 282001 (Other: IRAS); A28890 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2020-06-24; First posted 2020-09-16 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; olaparib; AZD1390; ceralasertib; AZD5305; durvalumab

STUDY DESIGN:
Intervention Model Description: The trial is designed as a randomised Phase I dose escalation platform study, using the TiTE CRM design to find the RP2D of each DDRi with RT combination. At the time of patient identification the treating centre will be informed of the allocated study arm following a pre-specified prioritisation schedule. Consenting participants will be randomised between DDRi with RT or RT only. Patients are not randomised between experimental arms nor will endpoints be compared between experimental arms. RT only participants will be pooled across the platform to provide contemporary data on toxicity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Radiotherapy only (Active Comparator)
  Interventions: Radiation: Radiotherapy
- Olaparib + radiotherapy (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: Olaparib Oral Tablet [Lynparza]
- AZD1390 + radiotherapy (Experimental)
  Interventions: Radiation: Radiotherapy; Drug: AZD1390
- Ceralasertib (AZD6738) + radiotherapy + Consolidation durvalumab (Experimental): This study arm will include up to 12 months of consolidation durvalumab for eligible participants following the completion of radiotherapy +/- DDRi.
  Interventions: Radiation: Radiotherapy; Drug: Ceralasertib; Drug: Durvalumab
- AZD5305 + radiotherapy + Consolidation durvalumab (Experimental): This study arm will include up to 12 months of consolidation durvalumab for eligible participants following the completion of radiotherapy +/- DDRi.
  Interventions: Radiation: Radiotherapy; Drug: AZD5305; Drug: Durvalumab
- RT + consolidation durvalumab (Active Comparator)
  Interventions: Radiation: Radiotherapy; Drug: Durvalumab
- Arm D - did not proceed (Experimental): Arm D - did not proceed
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Administered as 30 fractions of 2Gy. Total 60 60Gy. Administered once daily monday to friday.
Drug: Olaparib Oral Tablet [Lynparza] — Oral tablet
  Other Names: AZD2281
  Arms: Olaparib + radiotherapy
Drug: AZD1390 — Oral tablet
  Arms: AZD1390 + radiotherapy
Drug: Ceralasertib — Oral Tablet
  Other Names: AZD6738
  Arms: Ceralasertib (AZD6738) + radiotherapy + Consolidation durvalumab
Drug: AZD5305 — Oral Tablet
  Arms: AZD5305 + radiotherapy + Consolidation durvalumab
Drug: Durvalumab — 1500mg iv infusion
  Arms: AZD5305 + radiotherapy + Consolidation durvalumab; Ceralasertib (AZD6738) + radiotherapy + Consolidation durvalumab; RT + consolidation durvalumab

SUMMARY:
CONCORDE is a multi-institution, multi-arm, Phase IB study that will determine the recommended phase II dose (RP2D) and safety profiles of different DNA damage repair inhibitors (DDRis) when given in an open label fashion in combination with fixed dose curative intent radiotherapy (RT) in patients with stage IIB/IIIA/IIIB NSCLC, followed by up to 12 months of consolidation durvalumab immunotherapy in selected study arms. The RP2D will be evaluated by incorporating the number of observed dose limiting toxicities (DLTs) into a time to event continuous reassessment method (TiTE- CRM) model within each of the experimental arms. TiTE-CRM is used here to take into account longer-term toxicities up to 13.5 months post start of radiotherapy and use these to inform dose escalation decision making.

DETAILED DESCRIPTION:
Radiotherapy is an effective treatment for patients with non-small cell lung cancer (NSCLC) that has not spread beyond the chest area. Radiotherapy is used as a curative treatment but unfortunately for most patients the cancer can return. Radiotherapy kills cells by damaging their DNA. Cells have the ability to repair that damage, especially the cells of normal tissue. If DNA repair can be prevented radiotherapy should be more effective causing the cancer cells to die.

The study will use new drugs that affect how cells repair DNA damage, called DNA damage response inhibitors (DDRi). These will be given together with radiotherapy to hopefully improve the effectiveness of radiotherapy, followed by up to 12 months of durvalumab immunotherapy in selected study arms to develop the trial in line with the standard of care for NSCLC. The study will try to find out the most effective and safe dose of this combination treatment. This will be a clinical trial where patients due to have radiotherapy, with the hope of successful treatment that could lead to cure from their cancer or extension of life, will be offered entry onto the study. All patients will receive their radiotherapy, with 3 out of every 4 people also receiving a single DDRi drug alongside this. Both patients and study doctors will know prior to the start of the actual treatment whether a DDRi will be given, and if so which one; no placebos will be used. The patients will be followed closely to check for side effects and to assess how their cancer is responding to treatment. Blood samples will be taken to monitor treatment progress and to try to predict which patients are most likely to benefit from this type of combined treatment.

ELIGIBILITY:
Core Inclusion Criteria (Radiation Phase)

1. Histologically or cytologically confirmed NSCLC (patients where the local MDT agree the diagnosis is NSCLC after review of the available pathology and imaging at MDT can be enrolled after discussion with the CI).
2. Not suitable for concurrent chemoradiotherapy/surgery due to tumour or patient factors
3. Stage IIB and III (TNM 8th Edition).
4. Planned to receive RT at curative intent doses (i.e., 60Gy) as part of treatment plan (either with or without induction chemotherapy).
5. Patient considered suitable for radical RT by the local lung cancer multidisciplinary team and a clinical oncologist.
6. If chemotherapy has been given previously, the maximum interval between the last day of chemotherapy and the start of RT <10 weeks.
7. Age ≥18
8. Life expectancy estimated to be greater than 6 months.
9. Karnofsky Performance status ≥70.
10. MRC dyspnoea score <3.
11. Forced expiratory volume in one second (FEV1) ≥35% predicted and diffusing capacity of the lungs for carbon monoxide (DLCO or TLCO) ≥35% predicted.
12. Patient must be fully informed about the study and have signed the informed consent form.
13. Patient must be willing and able to comply with the protocol, have mental capacity and (if relevant) use effective contraception throughout treatment and for 4 months for women of childbearing potential, and 6 months for men after treatment completion. Treatment is defined as including the last dose of durvalumab or DDRi in the consolidation phase.
14. Adequate organ function as defined in master protocol.
15. Patient has a body weight of >30kg.

Core Exclusion Criteria (Radiation Phase)

1. Mixed non-small cell and small cell tumours.
2. Confirmed progressive disease during induction chemotherapy.
3. Participation in a study of an investigational agent or using an investigational device within 4 weeks prior to the anticipated start of treatment.
4. Current or previous malignant disease which may impact on a patient's estimated life expectancy (other than NSCLC).
5. History of interstitial pneumonitis.
6. Prior thoracic radiotherapy.
7. Prior treatment with pneumotoxic drugs, e.g. busulfan, bleomycin, within the past year. If prior therapy in lifetime, then exclude if history of pulmonary toxicities from administration. Patients who have received treatment with nitrosoureas (e.g., carmustine, lomustine) in the year before study entry without experiencing lung toxicity are allowed on study.
8. Mean resting corrected QT interval (QTcF) >470 msec obtained from 3 electrocardiograms.
9. Received a prior autologous or allogeneic organ or tissue transplantation.
10. Patients unable to swallow orally administered medications or chronic gastrointestinal (GI) disease likely to interfere with absorption of IMP in the opinion of the treating investigator (e.g. malabsorption syndrome, resection of the small bowel, poorly controlled inflammatory bowel disease etc.).
11. Grade 2 or higher peripheral sensory neuropathy.
12. Known positive test for human immunodeficiency virus, active hepatitis B or C infection.
13. Positive pregnancy test (at eligibility assessment for women of childbearing potential) or breast-feeding women.
14. Patients with persistent toxicities (>CTCAE grade 2) caused by previous cancer therapy, excluding alopecia.
15. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML) or with features suggestive of MDS/AML.
16. Major surgery within 2 weeks of confirmation of eligibility.
17. Patients considered a poor medical risk by the investigator due to a serious, uncontrolled medical disorder, non-malignant system disease or active uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, uncontrolled hypertension, uncontrolled atrial fibrillation, active bleeding, recent (within 3 months) myocardial infarction, major seizure, active COVID-19, any psychiatric disorder that prohibits obtaining informed consent.
18. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.
19. Exclusions as described in the relevant study arm protocol. Patients ineligible for a particular study arm may be considered for entry into an alternative study arm if an appropriate slot is available and they meet all the inclusion and exclusion criteria for that arm. This will need to be discussed with CTRU and the patient will be required to reconsent using the appropriate study arm PIS/ICF.

Core Inclusion Criteria (Consolidation Phase)

1. A minimum of 4 and a maximum of 8 weeks* have elapsed following completion of RT
2. Any toxicities from RT have resolved to grade 1. If patient has pneumonitis following RT treatment, this must be asymptomatic (grade 1). If pneumonitis is ≥2 or requiring steroids, then participant is not eligible
3. Karnofsky Performance status ≥70
4. The laboratory requirements set out in Table 1 of the master protocol are met
5. Patient has no known hypersensitivity to the excipients of durvalumab
6. Patient has body weight of >30kg *Investigators should ideally aim to start consolidation treatment within 6 weeks, following the receipt of the CT scan results to rule out progression.

Core Exclusion Criteria (Consolidation Phase)

1. Progressive disease during RT or at the end of RT treatment response assessment.
2. Participant declines treatment in the consolidation phase.
3. Patients who have received prior anti-PD-1 or anti PD-L1 treatment.
4. Major surgery within 4 weeks of confirmation of eligibility for consolidation phase.
5. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.
6. Patients considered a poor medical risk by the investigator due to a serious, uncontrolled medical disorder, non-malignant system disease, active GI infection or active uncontrolled infection.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease e.g., colitis or Crohn's disease), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-03-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Dose limiting Toxicities | 13.5 months after start of radiotherapy
  Dose-limiting toxicities (DLTs), within 13.5 months of starting radiotherapy, in order to establish the Recommended Phase II Dose (RP2D) of each DDRi-RT combination.

SECONDARY OUTCOMES:
Safety and toxicity | 2 years after end of RT
  Safety will be reported based on the occurrence of SAEs, SARs and SUSARs. Toxicity will be reported based on adverse events, as graded by CTCAE V5.0, and determined by routine clinical assessments at each centre.
Treatment compliance | End of trial treatment (DDRi and RT)
  Treatment compliance will be measured by overall radiotherapy treatment time and delays, omissions and reductions to treatment doses (both DDRi and RT).
Best overall response | 2 years after end of RT
  Best overall response will be measured as the best response (complete response, partial response or stable disease) recorded until disease progression, reported up to 2 years post-RT. This will be assessed using RECIST 1.1
Disease control | 2 years after end of RT
  This will be assessed using the Green Criteria. Disease Control includes either the complete disappearance of all evidence of malignant disease or residual radiographic abnormalities assessed by chest CT scan at 3 and 6 months after completion of RT, which then remains stable for an additional 6 months or more and which then qualifies as controlled local disease.
Progression-free survival | 2 years post-RT
  Participants who have not progressed at the time of analysis will be censored at the last date they were known to be alive and progression free
Overall survival | 2 years post-RT
  Participants who have not died at the time of analysis will be censored at the last date they were known to be alive
Changes in Health Related Quality of Life | 2 years after end of RT
  Health Related Quality of Life will be determined using EORTC QLQ-C30, IL-73 and IL-74
Objective response rate | 2 years after end of RT
  Objective response rate (ORR) is defined as the proportion of patients who have a partial or complete response to therapy. The proportion of patients with evaluable scans that achieve at least a partial response, as defined by RECIST v1.1(31), will be presented with 95% confidence intervals.
Changes in tumour size during and following treatment with DDRi-RT compared to RT alone. | 2 years after end of RT

OTHER OUTCOMES:
Assessment of mutations in components of DDR pathway in archival tumour and cfDNA prior to therapy | 2 years after end of RT
  Exploratory endpoint
Assessment of T cells within the archival tumour specimens | 2 years after end of RT
  Exploratory endpoint
Changes in cfDNA during and following treatment with DDRi-RT compared to RT alone. | 2 years after end of RT
  Exploratory endpoint
Changes in circulating biomarkers of cardiac and respiratory toxicity during and following treatment with DDRi-RT compared to RT alone. | 3 months post end of RT
  Exploratory endpoint
Changes in circulating peripheral T cell sub-sets during and following treatment with DDRi-RT compared to RT alone. | 2 years after end of RT
  Exploratory endpoint
Changes in lung parenchyma during and following treatment with DDRi-RT compared to RT alone. | 2 years after end of RT
  Exploratory endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Alastair Greystoke, MB ChB, MSc, PhD, Principal Investigator — Newcastle University; Corinne Faivre-Finn, MD, PhD, Principal Investigator — University of Manchester
Locations (14):
- United Kingdom (14):
  - Belfast City Hospital, Belfast
  - Birmingham Heartlands Hospital, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - The Royal Marsden Hospital Chelsea, Chelsea
  - Western General Hospital, Edinburgh
  - St James's University Hospital, Leeds
  - The Clatterbridge Cancer Centre, Liverpool
  - St Bartholomew's Hospitals, London
  - University College Hospital London, London
  - The Christie NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne Hospitals NHS Trust, Newcastle upon Tyne
  - Weston Park Hospital, Sheffield
  - The Royal Marsden Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data datasets generated and/or analysed during the current study will be available upon request from the Clinical Trials Research Unit, University of Leeds. Data will be made available at the end of the trial. Data will remain available from then on for as long as CTRU retains the data.
  CTRU makes data available by a 'controlled access' approach. Data will only be released for legitimate secondary research purposes, where the Chief Investigator, Sponsor and CTRU agree that the proposed use has scientific value and will be carried out to a high standard (in terms of scientific rigour and information governance and security), and that there are resources available to satisfy the request. Data will only be released in line with participants' consent, all applicable laws relating to data protection and confidentiality, and any contractual obligations to which the CTRU is subject.
Time Frame: At the end of the trial, i.e. usually when all primary and secondary endpoints have been met and all key analyses are complete.
Access Criteria: Contact CTRU-DataAccess@leeds.ac.uk in the first instance.
  No individual participant data will be released before an appropriate agreement is in place setting out the conditions of release. The agreement will govern data retention, usually stipulating that data recipients must delete their copy of the released data at the end of the planned project.
  The CTRU encourages a collaborative approach to data sharing, and believe it is best practice for researchers who generated datasets to be involved in subsequent uses of those datasets. Recipients of trial data for secondary research will also receive data dictionaries, copies of key trial documents and any other information required to understand and reuse the released datasets.
  The conditions of release for aggregate data may differ from those applying to individual participant data. Requests for aggregate data should also be sent to the above email address to discuss and agree suitable requirements for release.

REFERENCES:
- [Background] Faivre-Finn C, Brown S, Ryan A, Greystoke A; CONCORDE Investigators. The UK at the Forefront of Innovative Drug-Radiotherapy Combination Clinical Trials: Introducing the CONCORDE Platform. Clin Oncol (R Coll Radiol). 2020 Jun;32(6):358-362. doi: 10.1016/j.clon.2020.02.003. Epub 2020 Feb 24. No abstract available. PMID 32107107
- [Background] Walls GM, Oughton JB, Chalmers AJ, Brown S, Collinson F, Forster MD, Franks KN, Gilbert A, Hanna GG, Hannaway N, Harrow S, Haswell T, Hiley CT, Hinsley S, Krebs M, Murden G, Phillip R, Ryan AJ, Salem A, Sebag-Montefoire D, Shaw P, Twelves CJ, Walker K, Young RJ, Faivre-Finn C, Greystoke A. CONCORDE: A phase I platform study of novel agents in combination with conventional radiotherapy in non-small-cell lung cancer. Clin Transl Radiat Oncol. 2020 Sep 22;25:61-66. doi: 10.1016/j.ctro.2020.09.006. eCollection 2020 Nov. PMID 33072895
- [Derived] Walker K, Hinsley S, Phillip R, Oughton JB, Murden G, Chalmers AJ, Faivre-Finn C, Greystoke A, Brown SR; CONCORDE Investigators. Implementation of the Time-to-Event Continuous Reassessment Method Design in a Phase I Platform Trial Testing Novel Radiotherapy-Drug Combinations-CONCORDE. JCO Precis Oncol. 2022 Nov;6:e2200133. doi: 10.1200/PO.22.00133. PMID 36446040